CLINICAL TRIAL: NCT05791799
Title: A Multicenter Prospective Randomized Controlled Clinical Study of Etonogestrel Implants to Protect Ovarian Reserve Function in Systemic Lupus Erythematosus
Brief Title: Etonogestrel Implants Protect Ovarian Reserve Function in Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022ZSLYEC-461
Record Dates: First submitted 2023-02-01; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — etonogestrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etonogestrel implants group (Experimental): Women will be subjected to etonogestrel implant (68mg) insertion.
  Interventions: Drug: Etonogestrel
- control group (No Intervention): This group of women will not be intervened.

INTERVENTIONS:
Drug: Etonogestrel — Etongestrel implant will be implanted subcutaneously in the participant's non-dominant arm for one year
  Arms: Etonogestrel implants group

SUMMARY:
This clinical trial aims to test in female patients with systemic lupus erythematosus (SLE). The main question it seeks to answer is whether etonogestrel implants can protect ovarian reserve function in patients with SLE. Participants will be randomly divided into a test group and a control group. The test group will be implanted subcutaneously with etongestrel for one year. Researchers won't intervene in the control group. After three months of drug-eluting, researchers will compare measures of ovarian reserve function in the test and control groups to see if etonogestrel implants can protect ovarian reserve function in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Systemic lupus erythematosus was confirmed
2. 18-37 years old

Exclusion Criteria:

1. History of sex chromosome abnormalities
2. History of abnormal thyroid function
3. History of abnormal adrenal function
4. History of pituitary disease
5. History of sexual hormone drug use in the past 3 months
6. History of ovarian tumors or invasive ovarian operations
7. Pregnancy
8. Have a birth plan in the next 1 year
9. Ovarian failure

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian hormone (AMH) serum level | one year and three months
  The serum AMH levels of the two groups will be compared one year and three months after enrollment.

SECONDARY OUTCOMES:
Number of antral follicle | one year and three months
  The number of antral follicles will be recorded by transvaginal ultrasound and compared one year and three months after enrollment.
Follicle-stimulating hormone (FSH) serum level | one year and three months
  The serum FSH levels of the two groups will be compared one year and three months after enrollment.
luteinizing hormone (LH) serum level | one year and three months
  The serum LH levels of the two groups will be compared one year and three months after enrollment.
Estradiol (E2) serum level | one year and three months
  The serum E2 levels of the two groups will be compared one year and three months after enrollment.